CLINICAL TRIAL: NCT02635568
Title: Duration of Marijuana Concentration in Breast Milk- A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 15-1639
Record Dates: First submitted 2015-12-14; First posted 2015-12-21 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Cannabis; Pregnancy; Breast Feeding
MeSH Terms: conditions — Marijuana Abuse; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal breast milk, maternal urine, maternal plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cannabis Use — Observational Study

SUMMARY:
Legalization of marijuana in Colorado for both medicinal and recreational purposes has led to a perception of its safety, which has not been well studied in pregnant or lactating women. The psychoactive component of marijuana, delta-9-tetrahydrocannabinol (THC) is lipophilic and therefore presumed to be secreted into breast milk. Additionally, the difference between modes of consumption (ie. smoked vs. edible) has not been well described in regards to THC concentration in breast milk. The purpose of this small pilot study is to describe the presence and duration of THC expression in breast milk among women who have evidence of THC exposure at the time of labor and delivery or within 72 hours of delivery. The researchers hypothesize that women with positive urine drug screen for THC within 72 hours of delivery may excrete THC in breast milk for a predicted period of time, and therefore the aim of this project is to determine timing to safely return to breastfeeding to decrease infant exposure to THC.

The specific aims are to determine in women who test positive for THC at delivery:

1. Determine length of time THC and metabolites are detected in breast milk of mothers who have a positive urine drug screen at the time of presentation for labor and delivery or within 72 hours of delivery.
2. Determine length of time THC and metabolites are detected in breast milk of mothers with postnatal exposure of either ingested or inhaled marijuana, to inform recommendations on when to safely return to breastfeeding.
3. Describe modes of marijuana consumption in women presenting for delivery and correlate with THC concentrations and persistence in breast milk.

DETAILED DESCRIPTION:
This prospective, observational pilot study will identify women within 72 hours of delivery who have a positive urine drug screen for THC and who intend to breastfeed. Eligibility will not be dependent upon the disposition of the infant, either discharged shortly after birth or infants with NICU admission. The study will last six weeks from the time of enrollment. Mothers who consent to participate will complete an in-person survey on marijuana use and exposure during pregnancy at study entry and weekly surveys of current marijuana use. Samples of maternal breast milk, maternal urine, and infant urine will be collected at least three times, but no more than five times during the week (Monday - Friday) during infant hospitalization, dependent on maternal availability. If the infant is discharged from the hospital, visits will occur twice weekly during out-patient clinic visits. The presence of marijuana will be measured by THC concentrations in maternal breast milk, maternal urine and maternal plasma, collected by research staff at each visit. the investigators will ask mothers to refrain from feeding their baby their breast milk for at least 2 weeks after last marijuana exposure, which currently is the minimum time period recommended by lactation consultants in UCH and CHCO Neonatal Intensive Care Units (NICU). If a NICU admitted infant is medically stable to tolerate enteral feedings, they are given feedings either by mouth or by nasogastric feeding tubes, of either expressed breast milk, donor breast milk, or formula. The researchers current practice for infants admitted to the NICU is to offer donor breast to infants whose mothers cannot provide their own breast milk, for numerous reasons. Mothers of infants who are not in the NICU would be encouraged to pump breast milk and dump, for 2 weeks after last THC exposure while using formula until returning to breastfeeding. As this issue is commonly encountered in our clinical practice, the investigators find that many mothers are committed to providing safe feedings to their infants after given education regarding concerns of THC impact on infant development. The time point to safely return to breast milk following THC exposure is unknown, and is a primary aim of this study.

There are numerous documented benefits to breast milk, especially in preterm infants however sufficient literature exists to question the safety of THC's effects on the developing brain which may also be particularly susceptible in prematurity. Due to these unknown and understudied but highly concerning effects, The researchers faculty Neonatology practice has agreed to the consensus of refraining from knowingly administering breast milk from mothers actively using THC. Exemptions do occur in certain clinical settings. If this occurs during a mother's study enrollment, subsequent samples would be marked appropriately and the analytical data will be carefully examined.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be identified in two ways:

  1. Standard of care urine toxicology screening at the time of delivery: Women who test positive for THC on a urine toxicology screening who intend to breastfeed will be recruited within 72 hours of delivery at University of Colorado Hospital (UCH) and mothers whose infants are admitted to Children's Hospital Colorado (CHCO) NICU.
  2. Volunteers: Patients of UCH prenatal OB clinics, postpartum unit, and in the UCH and CHCO NICUs .

Exclusion Criteria:

* Mothers who do not intend to breastfeed; mothers less than 18 years of age; mothers who have positive urine drug for other illicit drugs (cocaine, methamphetamines).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients who test positive for THC on a urine toxicology screening who intend to breastfeed will be recruited within 72 hours of delivery.
  2. Using direct-to-patient advertising, the investigators plan to advertise the study in the UCH prenatal clinics, postpartum unit, and in the UCH and CHCO NICUs with an IRB approved flyer. Patients who volunteer will submit a confidential urine sample to the research staff when they present for delivery at UCH, or within 72 hours after delivery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of marijuana concentration in breast milk after use during pregnancy | Breast milk collection 2-5 times weekly for 6 weeks
  Determine length of time THC and metabolites are detected in breast milk of mothers who have a positive urine drug screen at the time of presentation for labor and delivery or within 72 hours of delivery.

SECONDARY OUTCOMES:
Duration of marijuana concentration in breast milk after postnatal use | Breast milk collection 2-5 times weekly for 6 weeks
  Determine length of time THC and metabolites are detected in breast milk of mothers with postnatal exposure of either ingested or inhaled marijuana, to inform recommendations on when to safely return to breastfeeding.
Frequency of marijuana use among postpartum women | One time weekly for 6 weeks
  Using a weekly survey, investigators will collect patient-reported information about modes of marijuana use and frequency. This data will be correlated with THC concentrations and persistence in breast milk.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Wymore, MD, Principal Investigator — Children's Hospital Colorado, University of Colorado Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: Undecided